CLINICAL TRIAL: NCT05659524
Title: Nasal Outcomes Using Saline Irrigations After Endonasal Pituitary Surgery - The NOSE Trial
Brief Title: Nasal Outcomes Using Saline Irrigations After Endonasal Pituitary Surgery
Acronym: NOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lori Wood (Other)
Collaborators: Barrow Brain and Spine (Unknown)
Responsible Party: Sponsor-Investigator, Lori Wood, Operations Manager of Neurosurgery Research, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHX-20-500-189-30-12
Record Dates: First submitted 2021-11-29; First posted 2022-12-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pituitary Tumor
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter randomized single-blinded, intervention trial involving 70 patients from this site (140 treated patients total from all sites), undergoing endoscopic transsphenoidal surgery for pituitary lesions. The same cohort will simultaneously be used to evaluate the role of sinonasal irrigations in those patients who undergo nasoseptal flap reconstructive procedures as part of their treatment.
Who Masked: Care Provider
Masking Description: The study will be blinded to the Otolaryngologist involved in the study. The research team and the patient will not be blinded. The goal of blinding the Otolaryngologist is to minimize the bias in grading the Lund Kennedy endoscopic scores which are a subjective metric interpreted in the office setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal saline irrigation (Active Comparator): Patients randomized to standard postoperative nasal care with twice a day saline sinonasal irrigations
  Interventions: Other: Nasal saline irrigation
- No Intervention (No Intervention): Patients randomized to not performing saline sinonasal irrigations.

INTERVENTIONS:
Other: Nasal saline irrigation — The following nasal care recommendations have been approved by the study protocol committee for patients randomized to the treatment arm with saline irrigations:
  * Postoperative days 1 through 3: patients will administer saline spray (e.g., Ocean nasal spray) to both nostrils four times daily.
  * Postoperative day 3 to week 12: patients will begin twice daily sinus irrigation rinse (e.g., NeilMed Sinus Rinse). They will perform 240 mL sinus rinses BID. After day 30, patients will perform sinus irrigation as needed. If a patient is unable to tolerate nasal rinses, saline spray can be used as an alternative.
  Arms: Nasal saline irrigation

SUMMARY:
This is a prospective, single-blinded, multicenter study evaluating the benefit of sinonasal irrigations following endoscopic pituitary surgery. The goal of this study is to create practice changing guidelines with objective data highlighting the importance of irrigations on postoperative outcomes for pituitary surgery.

DETAILED DESCRIPTION:
This prospective study, coupled with the results of the recent POET study evaluating the role of antibiotics in postoperative outcomes for pituitary surgery, will guide physicians in the optimal management of patients following endoscopic pituitary surgery.

The investigator group has an established record of completing multicenter studies (e.g., POET, TRANSPHER) that have influenced clinical practice guidelines, raised the profile of Barrow in the pituitary and skull base community, and resulted in numerous peer-reviewed publications and awards.

ELIGIBILITY:
Inclusion criteria

1. Adult patient undergoing endoscopic surgery for resection of pituitary tumors

   * nonfunctioning adenoma
   * acromegaly
   * prolactinoma
   * Rathke's cleft cyst
2. Adults >18 and <85 years of age
3. English speaking and able to understand the ASK Nasal-12 and SNOT-22 scales
4. Free of any physical, mental, or medical condition which, in the opinion of the investigator, makes study participation inadvisable
5. Planned binostril surgical approach
6. Either with or without septal flap reconstruction
7. Either with or without septoplasty

Exclusion criteria

1. Active sinus infection
2. Allergic rhinitis
3. Asthma
4. Vascular or inflammatory disease
5. History of previous sinonasal surgery
6. Any subject who is unwilling or unable to sign informed consent for the study
7. Pregnancy
8. Incarcerated patients
9. Cushing's disease
10. History of chronic sinusitis
11. Extended approaches to the skull base
12. Active sinusitis
13. Nasal polyps
14. Concurrent antibiotics for another indication (i.e., urinary tract infection)
15. Immunodeficiency
16. History of radiation to the skull base

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in mean sinonasal quality of life | 12 weeks
  Difference in mean sinonasal quality of life between groups as determined by patient reported Sino-nasal Outcome Test (SNOT-22) scores at 4 weeks. SNOT-22 scoring can be completed during a clinic visit or by phone interview. It is critical that the follow-up times are standardized because symptoms improve with time. A reduction in SNOT-22 composite score is indicative of improvement in symptoms.

SECONDARY OUTCOMES:
Endoscopy findings | 12 weeks
  Postoperative nasal endoscopy findings of purulence, nasal crusting, polyps, and synechiae as estimated on the Endoscopic Appearances scale developed by Lund- Kennedy at 1 week, 4 weeks, and 12 weeks after surgery.
Sinonasal quality of life as determined by patient-reported Anterior Skull Base Nasal Inventory-12 (ASK Nasal-12) scores | 12 weeks
  Sinonasal quality of life as determined by patient-reported ASK Nasal-12 scores at
  1week, 2 weeks, 4 weeks, 8 weeks and 12 weeks after surgery.
Sinonasal quality of life as determined by Sinonasal Outcomes Test 22 (SNOT-22) | 12 weeks
  Sinonasal quality of life as determined by Sinonasal Outcomes Test 22 (SNOT-22) overall scores at 1week, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after surgery.
Sinonasal quality of life as determined by SNOT-22 rhinological subscale scores | 12 weeks
  Sinonasal quality of life as determined by SNOT-22 rhinological subscale scores at 1 week, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after surgery.
Sinonasal quality of life, as determined by Sinonasal Outcomes Test 22 (SNOT-22), of subgroups including septal flap reconstruction and no septal flap reconstruction. | 12 weeks
  Sinonasal quality of life, as determined by Sinonasal Outcomes Test 22 (SNOT-22), of subgroups including septal flap reconstruction and no septal flap reconstruction.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Study is IRB approved to share deidentified data outside of the institution, with presence of a valid data sharing agreement.